CLINICAL TRIAL: NCT03451175
Title: Reproductibility of Cystometry in Multiple Sclerosis Patient
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Head of Neuro-Urology Department, Tenon Hospital, Pierre and Marie Curie University
Other Study IDs: P. GREEN 0001
Record Dates: First submitted 2018-02-11; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Lower Urinary Tract Symptoms; Cystometry; Multiple Sclerosis; Overactive Bladder; Overactive Detrusor
Keywords: Overactive Detrusor; Multiple Sclerosis; Reproductibility; Cystometry
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Multiple Sclerosis; Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the reproductibility (quantitative and qualitative) of cystometry in mutiple sclerosis patients.

DETAILED DESCRIPTION:
Some studies have evaluated the reproductibility of urodynamics in women with stress incontinence, and demonstrated a poor reproductibility of urodynamic parameters for a part of the studies and a good reproductibility for the others. There is only three studies investigating the reproductibility of repeated cystometries in patients with overactive detrusor and neurogenic lower tract dysfunction. The most common etiology in these studies is spinal cord injury. Only one article includes MS patients with lower urinary tract symptoms (22 patients among 226 with other etiologies).

The aim of this study was to assess the short term reproductibility in multiple sclerosis patients with qualitative and quantitative urodynamic data.

The authors conducted a prospective analysis in our Neuro-urology department of a University Hospital . All patient with Multiple Sclerosis referred for urinary disorders, coming for a urodynamic evaluation with multiple cystometries during the study were included if they had a detrusor overactivity for a filling of 300 ml or less on the first cystometry. The main exclusion criteria were a significate difference between the filling volume during the study and the volume truly of water truly collected after catheterization, an urinary tract infection, or an other acute disease.The investigators performed a first cystometry and looked for a detrusor overactivity, if the investigators discovered an involuntary detrusor contraction for a filling of 300 ml or less, the authors realized two others cystometries (filling rate of 50 mL/min) after informed consent. The volume and pressure at which the first and the maximal involuntary detrusor contraction, MCC were documented.

ELIGIBILITY:
Inclusion Criteria:

* All patient with Multiple Sclerosis referred for urinary disorders,
* coming for a urodynamic evaluation with multiple cystometries during the study - detrusor overactivity for a filling of 300 ml or less on the first cystometry.

Exclusion Criteria:

* significate difference between the filling volume during the study and the volume truly of water truly collected after catheterization,
* an urinary tract infection,
* an other acute disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis patients with overactive detrusor consulting in neurobiology center.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-07-02 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Reproductibility of urodynamic Capacity Cystometric Maximum (CCM) | 1 Day : during the urodynamic assessment
  Reproductibility of Capacity cystometric maximum (in ml) in the three cystometries evaluated using an intra class correlation
Reproductibility of urodynamic : Pressure maximum | 1 Day : during the urodynamic assessment
  Reproductibility of Pressure Maximum (in cmH2O) in the three cystometries evaluated using an intra class correlation
Reproductibility of urodynamic : Pressure of the first involuntary detrusor contraction (IDC) | 1 Day : during the urodynamic assessment
  Reproductibility of pressure of the first involuntary detrusor contraction (in cmH2O) in the three cystometries evaluated using an intra class correlation
Reproductibility of urodynamic : volume of filling for the first IDC | 1 Day : during the urodynamic assessment
  Reproductibility of volume of filling for the first involuntary detrusor contraction (in cmH2O) in the three cystometries evaluated using an intra class correlation

SECONDARY OUTCOMES:
Comparaison of urodynamic parameters between naive treatment patient and non naive treatment patients | 1 Day : during the urodynamic assessment
  Comparaison urodynamic parameters (CCM, Maximum pressure, volume filling of the first IDC, pressure of the first IDC) using a T student test

CONTACTS AND LOCATIONS:
Overall Officials: Gerard AMARENCO, PhD, Principal Investigator — GREEN GRC-01, Neuro-urology, hôpital Tenon
Locations (1):
- Service de Neuro-urology, hôpital Tenon, Paris, France